CLINICAL TRIAL: NCT03889093
Title: Radioembolization of Primary and Secondary Liver Malignancies and The Effect On The Immune System: A Prospective Study of Cytokine Modulation And Immune Cell Infiltration
Brief Title: Radioembolization of Primary and Secondary Liver Malignancies and The Effect On The Immune System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left Institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018LS026
Record Dates: First submitted 2019-03-12; First posted 2019-03-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Secondary Malignant Neoplasm of Liver
Keywords: peripheral blood monocytes; cytokine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Yttrium-90

STUDY DESIGN:
Intervention Model Description: Single arm prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yttrium-90 (Other): This single arm study is to evaluate immunologic changes following the treatment of primary or secondary malignancies of the liver utilizing beta-emitting, Yttrium-90.
  Interventions: Other: Yttrium-90

INTERVENTIONS:
Other: Yttrium-90 — This is to evaluate the immunologic effects of yttrium 90.

SUMMARY:
The goal of this study is to understand the immunologic effects radioembolization has on the immune system. This will be done by evaluating the changes on biopsy, peripheral blood monocytes, and cytokines.

DETAILED DESCRIPTION:
This is a single institution non-interventional study designed to evaluate the immune reaction to radioembolization (RE) of primary and secondary malignancies of the liver.

RE has been established as a standard of care treatment for both primary and secondary cancers of the liver. The treatment consists of a mapping, or planning angiogram, followed by a delivery angiogram where the dose of yttrium 90 (y90) is delivered. Data has been published on the immune modification powers of external beam radiation (XRT). However, very little data is available on the ways in which RE modifies the immune system. The goal of this study is to determine changes in the peripheral blood monocytes, cytokines and the treated and untreated liver tumors through sample collection prior to and for 12 weeks after standard of care RE.

The prior to, the RE delivery procedure patients will have a blood draw to evaluate for levels of 11 immunologically relevant cytokines (IL-1α, IL-1β, IL-2, IL-6, IL-10, IL-12p70, IL-18, TNFα, IFN-ϒ, Fit ligand 3, and MCP-1). These blood draws will be repeated at 7 days (- 2 days, + 5 days), 4 weeks (± 2 weeks) and 12 weeks (± 2 weeks) after RE.

The patients will also have the infiltration of immune relative cells into treated tumors evaluated. This will be done by the patients undergoing biopsy of the largest tumor to be treated prior to treatment and at 2 weeks (±7 days) following RE. If patients have other areas of tumor, which are not included in the initial treatment site, these areas will also be biopsied.

Finally, the change in immunologically important peripheral lymphocytes will be collected. This will be done with a blood draw on the day of, but prior to RE serving as an internal control. Patients will then also have blood draws performed at 7 days (±2 days), 4 weeks (± 2 weeks) and 12 weeks (± 2 weeks) after RE.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy or image (in the setting of hepatocellular carcinoma (HCC)) diagnosed hepatic malignancy
* Total bilirubin < 2 mg/dL
* ECOG status ≤ 2
* Life expectancy >3 months as documented in the medical record by the enrolling physician
* Age >22 years
* Lesion >2.0 cm which is amenable to percutaneously biopsied

Exclusion Criteria:

* Unwilling or unable to attend all study related follow ups
* Technetium 99 macro aggregated albumin (MAA) lung shunt fraction >20%
* Arterial anatomy which precludes the ability to safely perform RE
* INR > 1.8 or platelet count <50,000 which cannot be corrected
* Patients who are unable to hold anticoagulation and/or antiplatelet therapy in the periprocedural setting

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Change in concentrations of PBMC | 12 weeks
  Determine changes in the peripheral blood lymphocytes utilizing flow cytometery after radioembolization (RE) therapy for primary and secondary malignancies of the liver at 12 weeks.

SECONDARY OUTCOMES:
Change in concentrations of cytokines | 1, 4, 12 weeks
  Determine changes in the peripheral blood cytokines after radioembolization (RE) therapy for primary and secondary malignancies of the liver. Specifically cytokines IL-1α units/mg, IL-1β units/mg, IL-2 units/mg, IL-6 units/mg, IL-10 units/mg, IL-12p70 units/mg, IL-18 units/mg, TNFα units/mg, IFN-Y units/mg, Fit ligand 3 units/mg, and MCP-1 units/mg will be measured.
Change in concentrations of immune cell infiltration into the tumor | 1, 4, 12 weeks
  Determine the changes in infiltrating immune cells within the treated tumor, which occur after radioembolization (RE) therapy for primary and secondary malignancies of the liver. This will be accomplished by obtaining tissue samples of the treated tumor before and after treatment, then performing staining and cell counts to determine the change in cytotoxic t cells, t helper cells, natural kill cells, macrophages, and dendritic cells.
Change in concentrations of PBMC | 1 and 4 weeks
  Determine changes in the peripheral blood lymphocytes utilizing flow cytometery after radioembolization (RE) therapy for primary and secondary malignancies of the liver at 1 and 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Shamar J Young, Young, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03889093/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03889093/ICF_001.pdf